CLINICAL TRIAL: NCT06671301
Title: The Impact of Lifestyle Medicine on the Sense of Coherence and the Biological Age, in a Community Sample.
Brief Title: The Impact of Lifestyle Medicine on the Sense Of Coherence and Biological Age in a Community Sample
Acronym: PSAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Evelina Tamiolaki, Principal investigator, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2401
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers Only; Healthy Adults
Keywords: Stress; Lifestyle medicine; Telomeres; Sense of Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSAI group (Experimental): Behavioural counselling
  Interventions: Behavioral: PSAI
- Control group (Other): No intervention used
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: PSAI — Holistic stress management program implementing the pillars of Lifestyle Medicine
  Arms: PSAI group
Other: Usual Care — Usual care without specific treatment
  Arms: Control group

SUMMARY:
This two-arm, pilot, cross-over randomized controlled trial took place at Diabetes Laboratory, First Department of Propaedeutic Internal Medicine, Laikon General Hospital, School of Medicine, National and Kapodistrian University of Athens, Athens, Greece the from February 2024 to June of 2024. The study protocol was approved by the Ethics Committee of First Department of Propaedeutic Internal Medicine, Laiko General Hospital(Protocol no 2401/February 27,2024)and was consistent with the Helsinki Declaration for human studies.

DETAILED DESCRIPTION:
Pythagorean Self-Awareness Intervention (PSAI) to a sample of community volunteers without pre-existing pathology, with the aim of evaluating the effectiveness of PSAI compared to a control group. Primary goals are to improve lifestyle (6 pillars), increase sense of coherence, improve telomere length and reduce perceived stress. Secondary goals are to reduce negative emotions, fatigue, neuroticism and inflammation. Also, the increase in self-efficacy, emotional intelligence, health locus of control, satisfaction with life and finally the improvement of memory and blood pressure. Measurements will take place in both groups before and after the intervention and included: Self-report questionnaires for measuring psychometric and lifestyle factors, cognitive assessment, body measurements, hair cortisol concentrations and blood sampling for telomere length.

ELIGIBILITY:
Inclusion Criteria:

* Clinically healthy adults
* Speaking and writing in Greek language

Exclusion Criteria:

* Participation in another stress management trial
* diagnosis of any serious mental disorder
* short-term or long-term treatment with corticosteroids
* drug addiction

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Telomeres length | Before and after the intervention(2 months)
  Quantitative PCR (qPCR) to determine relative telomere length
Sense of Coherence | Before and after the intervention(2 months)
  Sense of Coherence was assessed with the Sense of Coherence scale (SOC-13). The scale consists of 13 items rated from 0 to 7. It is considered to have high internal consistency reliability and high validity when compared to other scales measuring the same personality trait.

SECONDARY OUTCOMES:
Perceived Stress Scale-14 | Before and after the intervention(2 months)
  To assess perceived stress, the Greek version of the PSS questionnaire was administered, which consists of 14 items, each graded on a 5-point Likert scale. More specifically, there are seven positive and seven negative items and the total score ranges from 0 to 56. Higher PSS scores indicate higher levels of perceived in the past month
Pittsburgh Sleep Quality Index | Before and after the intervention(2 months)
  Sleep quality was assessed using the Greek version of the PSQI questionnaire. The PSQI consists of 19 self-report questions, grouped into 7 components (subjective sense of sleep quality, awakening time, latent period, duration, usual sleep productivity, use of sleep medication and daytime dysfunction). The score ranges from 0 to 3, resulting in a total score ranging from 0=high sleep quality to 21=low sleep quality. A total score of > or = 5 indicates poor sleep
Med Diet Score | Before and after the intervention(2 months)
  The healthy lifestyle and self-monitoring questionnaire consists of 26 items, which are divided into a 4-point Likert scale ranging from 1=never/rarely to 4= always. A higher score indicates increased health empowerment. Specifically, the HLPCQ is designed to assess one's degree of control over daily activities such as diet, daily schedule, physical activity, socialization and pessimistic thoughts
Electrolytic Extracellular Bioimpedance Tomography (TomEEX) | Before and after the intervention(2 months)
  A non invasive diagnostic tool that assesses various body functions, including: (a) stress response, (b) sensory and autonomic tones and (c) activation of limbic and cortical regions of the brain. In addition, it measures sodium (Na+) and chloride (CI-) levels in 17 areas of the body.
Body composition analysis | Before and after the intervention(2 months)
  Body Impedance analyzer used to estimate body composition analysis and is based on the principles of bioelectrical impedance. Impedance was measured through the legs and lower torso through a metal plate which incorporated the electrodes, as subjects stood barefoot
Positive and Negative Affect Schedule | Before and after the intervention(2 months)
  a self-report instrument to assess two basic dimensions of mood: positive and negative affect. The given tool consists of two scales of 10 pieces. Each element refers to a different emotion. The respondent reports the extent to which they felt each of the emotions in the past week according to a 5-point Likert scale (1= very slightly or not at all, 5=extremely
General Efficacy Scale | Before and after the intervention(2 months)
  This metric assessed each individual's perception of their abilities to work through challenging conditions and overcome everyday obstacles. It is based on a 4-point Liker-type scale ranging from 1 (not at all true) to 4 (absolutely true). The overall result is calculated by the sum of all statements. The psychometric properties of the aforementioned tool seem to be good in the Greek population
Life Satisfaction | Before and after the intervention(2 months)
  consists of 15 questions and 5 self-report statements and assesses three dimensions: conscious, mental and critical evaluation of the person's life
Big Five Personality | Before and after the intervention(2 months)
  measures five personality dimensions: Openness to experience, Conscientiousness, Extraversion, Agreeableness and Neuroticism and enjoys high reliability. It consists of 44 items and the respondent is asked to indicate how much they agree or disagree with each statement, where 1=Strongly Disagree, 2= Slightly Disagree, 3= Neither Agree nor Disagree, 4= Strongly Agree
Wong and Low Emotional Intelligence Scale | Before and after the intervention(2 months)
  questions about how a person manages their emotions in general. The Wong-Low scale is the scale of emotional intelligence and is consists of 16 items and the participant is asked to grade gradually from 1 to 7, where the grade "1" expresses the absolute disagreement with the sentence and "7" the absolute agreement.
Brief international assessment of cognition | Before and after the intervention(2 months)
  The standardized battery (BICAMS) was used to assess cognitive functions in the participants. This memory assessment tool took about 15 minutes to complete is completed and included three categories of cognitive tests: The Normal Symbol Digital Modalities Test (SDMT), which measured information processing speed, the California Verbal Learning Test-II (CVLT-II), which assessed verbal memory and subsequent immediate recall. Finally, the third test concerned short visuospatial memory Test Revised (BVMTR), which assessed visual memory and immediate recall. Low scores indicated cognitive dysfunctions and cognitive decline. The specific tool for memory assessment has been proposed to help practitioners identify a potential cognitive dysfunction in humans

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaos Tentolouris, Professor, Study Director — First Department of Propaedeutic Internal Medicine, Medical School, NKUA, Greece
Locations (1):
- Post-graduate course of Stress Science and Health Promotion, NKUA, Athens, Greece

IPD SHARING:
Plan to Share IPD: No
Upon request

REFERENCES:
- [Background] Athanasopoulou S, Simos D, Charalampopoulou M, Tentolouris N, Kokkinos A, Bacopoulou F, Aggelopoulou E, Zigkiri E, Chrousos GP, Darviri C, Gonos ES. Significant improvement of stress and aging biomarkers using a novel stress management program with the cognitive restructuring method "Pythagorean Self-Awareness Intervention" in patients with type 2 diabetes mellitus and healthy adults. Mech Ageing Dev. 2021 Sep;198:111538. doi: 10.1016/j.mad.2021.111538. Epub 2021 Jul 1. PMID 34217756
- [Background] Zigkiri ES, Nicolaides NC, Bacopoulou F, Simos D, Vlachakis D, Chrousos GP, Darviri C. The Effect of the Pythagorean Self-Awareness Intervention on Psychological, Lifestyle and Cognitive Measures of a Community Sample. J Mol Biochem. 2020;9(1):32-40. Epub 2020 Dec 30. PMID 33520744
- [Background] Charalampopoulou M, Bacopoulou F, Syrigos KN, Filopoulos E, Chrousos GP, Darviri C. The effects of Pythagorean Self-Awareness Intervention on breast cancer patients undergoing adjuvant therapy: A pilot randomized controlled trial. Breast. 2020 Feb;49:210-218. doi: 10.1016/j.breast.2019.12.012. Epub 2019 Dec 20. PMID 31901782
- [Background] Simos DS, Kokkinos A, Tentolouris N, Dimosthenopoulos C, Mantzou E, Artemiadis A, Bacopoulou F, Nicolaides NC, Kosta O, Chrousos GP, Darviri C. Pythagorean self-awareness intervention: A novel cognitive stress management technique for body weight control. Eur J Clin Invest. 2019 Oct;49(10):e13164. doi: 10.1111/eci.13164. Epub 2019 Sep 16. PMID 31421060